CLINICAL TRIAL: NCT00061932
Title: A Phase II Study of PS-341 Alone or in Combination With Irinotecan in Patients With Adenocarcinoma of the Gastroesophageal Junction (GEJ) or Stomach
Brief Title: Bortezomib With or Without Irinotecan in Treating Patients With Cancer of the Gastroesophageal Junction or Stomach
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03015; N01CM62204 (NIH)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Diffuse Adenocarcinoma of the Stomach; Intestinal Adenocarcinoma of the Stomach; Mixed Adenocarcinoma of the Stomach; Recurrent Gastric Cancer; Stage IIIB Gastric Cancer; Stage IIIC Gastric Cancer; Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Bortezomib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stratum 1 (previously untreated) (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11 and irinotecan IV over 90 minutes on days 1 and 8.
  Interventions: Drug: bortezomib; Drug: irinotecan
- Stratum 2 (previously treated) (Experimental): (closed to accrual as of 9/19/2006): Patients receive bortezomib as in stratum 1.
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: irinotecan — Given IV
  Other Names: Campto; Camptosar; CPT-11; U-101440E
  Arms: Stratum 1 (previously untreated)

SUMMARY:
This phase II trial is studying how well bortezomib with or without irinotecan works in treating patients with gastroesophageal junction or stomach cancer that can not be removed by surgery. Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Drugs used in chemotherapy such as irinotecan use different ways to stop tumor cells from dividing so they stop growing or die. Combining bortezomib with irinotecan may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate for the combination of irinotecan and PS 341 in patients with previously untreated adenocarcinoma of the stomach or GEJ.

II. To determine the response rate for PS341 in patients with previously treated adenocarcinoma of the stomach or GEJ.

III. To determine the toxicities and recovery from toxicities for patients receiving PS 341 alone or in combination with irinotecan IV. To perform GeneChip analysis on biopsy specimens prior to and subsequent to treatment with PS341 to determine changes in patterns of gene expression

OUTLINE: Patients are stratified (stratum 2 closed to accrual as of 9/19/2006) according to prior chemotherapy for advanced disease (yes vs no).

STRATUM 1 (Previously untreated patients): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11 and irinotecan IV over 90 minutes on days 1 and 8.

STRATUM 2 (Previously treated patients) (closed to accrual as of 9/19/2006): Patients receive bortezomib as in stratum 1.

In both strata, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the GE junction or stomach, which is beyond the scope of surgical resection
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Patients may have received adjuvant therapy for resected disease

  * Patients who have received no prior systemic therapy for advanced disease are eligible to receive PS341 + irinotecan
  * Patients are eligible for PS-341 as a single agent if they have received any number of prior regimens for gastric cancer
* Life expectancy of greater than 6 weeks
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >=100,000/uL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits
* When possible, patients will undergo an esophagogastroduodenoscopy (EGD) with biopsy prior to therapy then at 24 hours after starting PS-341
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents, concurrent radiation therapy, or other chemotherapy; patients who have had photodynamic therapy either within 4 weeks of study entry or concurrently are ineligible, unless it was used to relieve esophageal obstruction that could not be treated with laser, stent or dilatation
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PS 341 or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with PS341
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study
* Patients with a concurrent malignancy are excluded (except for early stage squamous cell carcinoma of the skin or cervix which can be treated locally); patients with an advanced malignancy within the past five years are not eligible; patients with a prior malignancy who have been disease free for five years are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2003-04; Primary Completion 2009-12 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allyson Ocean, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Result] Ocean AJ, Christos P, Sparano JA, Shah MA, Yantiss RK, Cheng J, Lin J, Papetti M, Matulich D, Schnoll-Sussman F, Besanceney-Webler C, Xiang J, Ward M, Dilts KT, Keresztes R, Holloway S, Chen EX, Wright JJ, Lane ME. Phase II trial of bortezomib alone or in combination with irinotecan in patients with adenocarcinoma of the gastroesophageal junction or stomach. Invest New Drugs. 2014 Jun;32(3):542-8. doi: 10.1007/s10637-014-0070-0. Epub 2014 Feb 15. PMID 24526575

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 41 patients were enrolled from 6 institutions between April 2003 and September 2006
Groups:
- Stratum 1 (Previously Untreated): Patients receive bortezomib IV 1.3 mg/m2 over 3-5 seconds on days 1, 4, 8, and 11 and irinotecan IV 125 mg/m2 over 90 minutes on days 1 and 8.
  bortezomib: Given IV (1.3 mg/m2)
  irinotecan: Given IV (125 mg/m2)
- Stratum 2 (Previously Treated): (closed to accrual as of 9/19/2006): Patients receive bortezomib as in stratum 1.
  bortezomib: Given IV
  irinotecan: Given IV
Period: Overall Study
Arm/Group | Stratum 1 (Previously Untreated) | Stratum 2 (Previously Treated)
Started | 29 | 12
Completed | 16 | 8
Not Completed | 13 | 4
Not completed — Withdrawal by Subject | 13 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 (Previously Untreated) | Stratum 2 (Previously Treated) | Total
Number analyzed (Participants) | 29 | 12 | 41
Age, Continuous [Median (Full Range); unit: years] | 58.5 [33 to 87] | 54.5 [33 to 77] | 56.5 [33 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 22 | 5 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  White | 24 | 9 | 33
  Asian | 2 | 2 | 4
  Black | 3 | 0 | 3
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: True Response Rate Evaluated for the Combination of Irinotecan and PS341 by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: CT or MRI imaging scans of measurable lesions were obtained at baseline and every 8 weeks thereafter. Responses were classified according to RECIST criteria (version 1.0)
Time Frame: Up to 6 years
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Stratum 1 (Previously Untreated) | Stratum 2 (Previously Treated)
Number analyzed (Participants) | 29 | 12
participants | 3 [2.2 to 27.4] | 1 [.2 to 38.5]

2. Secondary Outcome: Change in Patterns of Gene Expression Pre- and Post-treatment Performed by GeneChip Analysis
Description: Number of Participants with a Change in Gene Expression from Pre to Post Treatment
Time Frame: Baseline to 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1 (Previously Untreated) | Stratum 2 (Previously Treated)
Number analyzed (Participants) | 10 | 2
Participants | 2 | 2

ADVERSE EVENTS:
Arm/Group | Stratum 1 (Previously Untreated) | Stratum 2 (Previously Treated)
Serious Adverse Events (participants affected / at risk) | 24/29 | 8/12
Other Adverse Events (participants affected / at risk) | 25/29 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 (Previously Untreated) (N=29) | Stratum 2 (Previously Treated) (N=12)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Leukocytopenia (Investigations) | 8 (8) | 0 (0)
Neutropenia (Investigations) | 8 (8) | 0 (0)
Thrombocytopenia (Investigations) | 3 (3) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Heart stoppage (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 5 (5) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Edema: trunk/genital (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (5) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Infection: Lung (Infections and infestations) | 0 (0) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Obstruction: Small bowel NOS (Gastrointestinal disorders) | 4 (4) | 1 (1)
Pain: right hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Rash: desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 (Previously Untreated) (N=29) | Stratum 2 (Previously Treated) (N=12)
Fever (in the absence of neutropenia) (General disorders) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 4 (4) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Neuropathy: Sensory (Nervous system disorders) | 4 (4) | 0 (0)
Chills (General disorders) | 4 (4) | 0 (0)
Edema:limbs (General disorders) | 4 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 5 (5)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Rash: desquamation (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less